CLINICAL TRIAL: NCT01042561
Title: Vitamin D Status and Dose Response in Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nebraska (Other)
Collaborators: Creighton University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 0281-09-FB
Record Dates: First submitted 2009-12-31; First posted 2010-01-05 (Estimated); Last update posted 2023-09-01 (Actual); Status verified 2023-08

CONDITIONS: Vitamin D; Prematurity
Keywords: vitamin d; prematurity; 25(OH)D; infant; CRP; PTH
MeSH Terms: conditions — Premature Birth | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator): This group will recieve the current standard of care for infants in the NICU, recieving infant formula that provides less than 400 IU of vitamin D a day.
  Interventions: Dietary Supplement: vitamin D3 placebo
- Vitamin D (Experimental): This group will recieve standard of care infant formulas that provide less than 400 IU of vitamin D a day, in addition they will be supplemented with 400 IU of vitamin D3 daily.
  Interventions: Dietary Supplement: Vitamin D3

INTERVENTIONS:
Dietary Supplement: Vitamin D3 — 400 IU of vitamin D3 daily. Pts will recieve 1 mL a day with a feeding for 28 days.
  Other Names: DVi-Sol
  Arms: Vitamin D
Dietary Supplement: vitamin D3 placebo — Placebo designed by research pharmacist. Pts will recieve 1 mL a day with feedings for 28 days.
  Arms: placebo

SUMMARY:
This study will examine the relationship of serum 25(OH)D levels in infants 32 weeks and greater gestation who are fed infant formula to markers of inflammation and bone metabolism.

DETAILED DESCRIPTION:
It is hypothesized that serum 25(OH)D levels in infants 32 weeks and greater gestation are not maintained at optimal levels of greater than 32 ng/Ml with currently available infant formulas, and that this will have an inverse relationship with markers of inflammation and bone metabolism.

ELIGIBILITY:
Inclusion Criteria:

* greater than 32 weeks gestation,
* exclusively formula fed.

Exclusion Criteria:

* less than 32 weeks gestation,
* less than 1500 grams,
* recieving maternal breast milk,
* recieving parenteral nutrition,
* congenital anomolies,
* disorders of vitamin D metabolism,
* inborn errors of metabolism,
* seizure disorders,
* parathroid disease,
* liver, GI tract, or kidney disease, and
* disorders of calcium metabolism.

Ages: 5 Minutes to 3 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 64 (Actual)
Dates: Start 2009-08-07 (Actual); Primary Completion 2010-08-01 (Actual); Study Completion 2010-08-01 (Actual)

PRIMARY OUTCOMES:
Serum 25-Hydroxyvitamin D [25(OH)D] Levels | 30 days
  Total serum 25(OH)D level is currently considered the best indicator of vitamin D supply to the body from cutaneous synthesis and nutritional intake. For infants, ≤37.5 nmol/L (15 ng/mL) would be considered indicative of deficiency and >50 nmol/L (20 ng/mL) as indicative of vitamin D sufficiency.

SECONDARY OUTCOMES:
Serum C-reactive protein (CRP) | 30 days
  Serum C-reactive protein (CRP) is a protein made by the liver and increases when there's inflammation in the body. The upper normal reference levels range from 6 to 20 mg/L as cutoff levels to indicate the presence of sepsis or infection.
Serum intact parathyroid hormone (iPTH) | 30 days
  Secretion of parathyroid hormone (PTH) is regulated by the level of calcium in the blood. Low serum calcium causes increased PTH to be secreted, whereas increased serum calcium inhibits PTH release. Normal values are 10 to 55 picograms per milliliter (pg/mL).

CONTACTS AND LOCATIONS:
Overall Officials: Corrine Hanson, PhD, RD, Principal Investigator — University of Nebraska
Locations (1):
- University of Nebraska Medical Center, Omaha, Nebraska, United States

REFERENCES:
- [Derived] Huey SL, Acharya N, Silver A, Sheni R, Yu EA, Pena-Rosas JP, Mehta S. Effects of oral vitamin D supplementation on linear growth and other health outcomes among children under five years of age. Cochrane Database Syst Rev. 2020 Dec 8;12(12):CD012875. doi: 10.1002/14651858.CD012875.pub2. PMID 33305842